CLINICAL TRIAL: NCT04801537
Title: Association of Temperature of Extremities and Necrotizing Enterocolitis(NEC)
Brief Title: Temperature of Extremities and Necrotizing Enterocolitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Collaborators: Children's Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Chen Long,MD, director, Children's Hospital of Chongqing Medical University
Other Study IDs: neutral temperature
Record Dates: First submitted 2021-03-12; First posted 2021-03-17 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Neutral Temperature; Bloody Stool; Necrotizing Enterocolitis
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Enterocolitis, Necrotizing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- normal body temperature and warm extremities: standard set of environmental temperature is done, and the infant's body temperature is normal and extremities are warm
  Interventions: Other: normal body temperature and warm extremities
- normal body temperature and cold extremities: standard set of environmental temperature is done, and infant's body temperature is normal and extremities are cold
  Interventions: Other: normal body temperature and cold extremities

INTERVENTIONS:
Other: normal body temperature and warm extremities — environmental temperature is set according to the standard method to keep normal body temperature and warm extremities
  Groups: normal body temperature and warm extremities
Other: normal body temperature and cold extremities — environmental temperature is set according to the standard method to keep normal body temperature, but cold extremities
  Groups: normal body temperature and cold extremities

SUMMARY:
Bloody stool and necrotizing enterocolitis(NEC) is two main focus in non-neonatal intensive care unit ward and usually lead to longed duration of hospitalization.

Neutral temperature is a environmental temperature where the infant's body temperature is normal under resting state, and the changes of body temperature and skin temperature are less than 0.2-0.3 centigrade. According the definition, a suggested temperature range is set. For example, if an infant's body weight is more than 2500 gram, the initial set of environmental temperature is 31.3 centigrade with a range of 29.8-32.8 centigrade.

low environmental temperature is a risk factor for Bloody stool and NEC. Therefore, how to set the optimal environmental temperature is a challenge.

DETAILED DESCRIPTION:
After birth, newborns must adapt to their relatively cold environment by the metabolic production of heat because they are not able to generate an adequate shivering response. Under the condition, environment temperature should be given to protect an infant from cold stress and cold injury, even NEC.

Therefore, the setting of the optimal environment temperature is a key focus in neonatal ward. Here, the investigators suggest a hypothesis that environment temperature should be set to keep warmth of extremities temperature and infant's body temperature is between 36.7-37.3 centigrade.

In the present study, the investigators will test the hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* body weight >2500 grams and/or gestational age >35 weeks
* an infant is diagnosed with hyperbilirubinemia and/or pneumonia without need for oxygen inhalation

Exclusion Criteria:

* congenital deformities
* refusal of parents' consent

Ages: 1 Hour to 28 Days | Sex: All
Age Groups: Child
Study Population: an infant's body weight > 2500 grams and/or gestational age >35 weeks is included in the present study.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
bloody stool | before discharge
  a infant is suffered from bloody stool
necrotizing entercolitis(NEC) | before discharge
  a infant is suffered from NEC

SECONDARY OUTCOMES:
late-onset sepsis(LOS) | before discharge
  a infant is suffered from LOS

CONTACTS AND LOCATIONS:
Locations (1):
- Chen, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided